CLINICAL TRIAL: NCT04853576
Title: A Phase 1/2 Study to Evaluate the Safety and Efficacy of a Single Dose of Autologous Clustered Regularly Interspaced Short Palindromic Repeats Gene-edited CD34+ Human Hematopoietic Stem and Progenitor Cells (EDIT-301) in Subjects With Severe Sickle Cell Disease
Brief Title: A Study Evaluating the Safety and Efficacy of EDIT-301 in Participants With Severe Sickle Cell Disease (RUBY)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Editas Medicine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EM-SCD-301-001
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Sickle Cell Disease; Hemoglobinopathies
Keywords: Anemia; Anemia, Sickle Cell; Anemia, Hemolytic, Congenital; Anemia, Hemolytic; Genetic Diseases, Inborn; Cell Disorders, Sickle; HbS Disease; Sickling Disorder Due to Hemoglobin S; Hematologic Diseases
MeSH Terms: conditions — Anemia, Sickle Cell; Hemoglobinopathies; Anemia; Anemia, Hemolytic, Congenital; Anemia, Hemolytic; Genetic Diseases, Inborn; Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EDIT-301 (Experimental): EDIT-301 (autologous gene edited (CD)34+ hematopoietic stem cells) will be administered as a one-time intravenous infusion.
  Interventions: Genetic: EDIT-301

INTERVENTIONS:
Genetic: EDIT-301 — Administered by IV infusion after myeloablative conditioning with busulfan.
  Other Names: renizgamglogene autogedtemcel; reni-cel

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of treatment with EDIT-301 in adult and adolescent participants with severe sickle cell disease (SCD).

DETAILED DESCRIPTION:
This is a Phase 1/2 single-arm, open-label, multicenter study evaluating the safety and efficacy of a single unit dose of EDIT-301 for autologous hematopoietic stem cell transplant (HSCT) in subjects with severe SCD. Planned study subjects will be comprised of male and female adult and adolescent subjects with severe SCD, from 12 to 50 years of age, inclusive.

ELIGIBILITY:
Key Inclusion Criteria:

Diagnosis of severe sickle cell disease as defined by:

* Documented SCD genotype (βS/βS, βS/β0, βS/β+, or others) and
* History of at least two severe vaso-occlusive events per year requiring medical attention despite hydroxyurea or other supportive care measures in the two year-period prior to provision of informed consent or assent, as applicable

Karnofsky (for subjects >16 years of age) or Lansky (for subjects ≤ 16 years of age) Performance Status ≥ 80%

Normal transcranial doppler velocity in subjects 16 years of age or younger

Key Exclusion Criteria:

* Available 10/10 HLA-matched related donor
* Prior HSCT or contraindications to autologous HSCT
* Any contraindications to the use of plerixafor during the mobilization of hematopoietic stem cells (HSCs) and any contraindications to the use of busulfan and any other medicinal products required during the myeloablative conditioning, including hypersensitivity to the active substances or to any of the excipients
* Unable to receive red blood cell (RBC) transfusion for any reason
* Unable or unwilling to comply with standard of care changes in background medical treatment in preparation of, during, or following HSCT, including and not limited to discontinuation of hydroxyurea, voxelotor, crizanlizumab, or L-glutamine
* Any history of severe cerebral vasculopathy
* Inadequate end organ function
* Advanced liver disease
* Any prior or current malignancy or immunodeficiency disorder
* Immediate family member with a known or suspected Familial Cancer Syndrome
* Clinically significant and active bacterial, viral, fungal, or parasitic infection

Other protocol defined inclusion/exclusion criteria may apply

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-05-04 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving complete resolution of severe vaso-occlusive events (VOEs) | from Month 6 through Month 18 post EDIT-301 infusion

SECONDARY OUTCOMES:
Proportion of subjects achieving complete resolution of VOEs | from Month 6 through Month 18 post EDIT-301 infusion
Proportion of subjects with 90% reduction in annualized rate of severe VOE compared to pre-treatment period | starting from 6 months up to 2 years post EDIT-301 infusion
Proportion of subjects with 75% reduction in annualized rate of severe VOE compared to pre-treatment period | starting from 6 months up to 2 years post EDIT-301 infusion
Proportion of subjects with 50% reduction in annualized rate of severe VOE compared to pre-treatment period | starting from 6 months up to 2 years post EDIT-301 infusion
Difference (pre-treatment vs. post-treatment) in annualized rates of severe VOEs | starting from 6 months up to 2 years post EDIT-301 infusion
Difference (pre-treatment vs. post-treatment) in annualized rate of hospitalization for severe VOEs | starting from 6 months up to 2 years post EDIT-301 infusion
Proportion of subjects with sustained HbF ≥ 20% (HbF/Hb) compared with baseline | starting from 6 months up to 2 years post EDIT-301 infusion
Proportion of subjects with mean HbF ≥ 30% (HbF/Hb) compared with baseline | starting from 6 months up to 2 years post EDIT-301 infusion
Proportion of subjects with mean total Hb ≥ 10 g/dL compared with baseline | starting from 6 months up to 2 years post EDIT-301 infusion
Proportion of subjects with mean total Hb increase from baseline of ≥ 2 g/dL | starting from 6 months up to 2 years post EDIT-301 infusion
Difference (pre-treatment versus post-treatment) in annualized number of units of pRBC transfused for SCD-related indications | starting from 6 months up to 2 years post EDIT-301 infusion
Change from baseline in HbF concentration (g/dL) | up to 2 years post EDIT-301 infusion
Change from baseline in total Hb concentration (g/dL) | up to 2 years post EDIT-301 infusion
Change from baseline in markers of hemolysis (absolute reticulocyte count, indirect bilirubin, lactate dehydrogenase, haptoglobin) | up to 2 years post EDIT-301 infusion
Time to neutrophil engraftment (the first day in which 3 consecutive absolute neutrophil count (ANC) ≥ 0.5 x 109/L laboratory values obtained on different days) | up to 24 months after EDIT-301 infusion
Time to platelet engraftment (the first day in which 3 consecutive platelets ≥ 50 x 109/L laboratory values obtained for at least 7 days following the last platelet transfusion and 10 days following any administration of thrombopoietin (TPO) mimetics) | up to 24 months after EDIT-301 infusion
Frequency and severity of adverse events (AEs) | up to 24 months post EDIT-301 infusion

CONTACTS AND LOCATIONS:
Locations (24):
- United States (21):
  - UCSF Benioff Children's Hospital, Oakland, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Smilow Cancer Hospital, New Haven, Connecticut
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University Medical Center - Department of Pediatrics, New York, New York
  - Columbia University Medical Center, New York, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Atrium Health, Charlotte, North Carolina
  - University Hospitals Rainbow Babies & Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The James Cancer Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Tristar Medical Group Children's Specialists/Sarah Cannon Center for Blood Cancers, Nashville, Tennessee
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Cook Children's, Fort Worth, Texas
- Canada (3):
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No